CLINICAL TRIAL: NCT00509431
Title: A Phase I/II, Dual-Center, Open-Label Trial of the Safety and Efficacy of Tarceva™ (Erlotinib Hydrochloride) Plus Sirolimus in Patients With Recurrent Malignant Glioma Not on P450-Inducing Anti-Epileptics
Brief Title: Erlotinib and Sirolimus in Treating Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000557423; UCLA-0604104
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2016-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult gliosarcoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; recurrent adult brain tumor; adult glioblastoma; adult pilocytic astrocytoma; adult diffuse astrocytoma; adult subependymal giant cell astrocytoma; adult oligodendroglioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Astrocytoma; Oligodendroglioma; Glioma; Brain Neoplasms | interventions — Erlotinib Hydrochloride; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib + Sirolimus (Experimental): This is an open-label,phase I single-arm dose-escalation and phase II study of continuous, once daily doses of erlotinib administered orally in combination with sirolimus in adult patients with malignant glioma at first, second or third recurrence
  Interventions: Drug: Erlotinib + Sirolimus

INTERVENTIONS:
Drug: Erlotinib + Sirolimus — In arm I of dose escalation phase,starting dose of erlotinib is 150 mg daily. Starting dose of sirolimus includes a 15 mg loading dose, followed by continuous dosing at 5 mg daily.Dose escalation will proceed according to protocol Phase II of the study was not conducted only Phase I

SUMMARY:
RATIONALE: Erlotinib and sirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I/II trial is studying the side effects and best dose of erlotinib when given together with sirolimus and to see how well they work in treating patients with recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of escalating doses of erlotinib hydrochloride in combination with sirolimus in adult patients with malignant glioma, who are not receiving enzyme-inducing anti-epileptic drugs (EIAED). (Phase I)
* Evaluate preliminary efficacy (response rate [RR], progression-free survival [PFS], and overall survival [OS]) of erlotinib hydrochloride and sirolimus combination therapy in glioblastoma multiforme (GMB)/gliosarcoma (GS) patients who are not undergoing surgery at the time of recurrence or relapse (dose-expansion arm). (Phase II)
* Evaluate molecular determinants of response to the combination of erlotinib hydrochloride and sirolimus, especially the roles of the mutation of EGFR (e.g., vIII mutant, other somatic mutations of vIII, and mutation/deletion of PTEN).

Secondary

* To characterize the safety and tolerability of erlotinib hydrochloride and sirolimus combination therapy in these patient populations.
* To characterize the single-dose and repeated-dose pharmacokinetic (PK) profiles of erlotinib hydrochloride (in serum) and sirolimus (in whole blood) combination therapy in these patient populations.
* To characterize, in pre- and/or post-treatment tumor samples, when available, expression levels of total and activated phosphorylated proteins relevant to the EGFR, VEGFR, and PI3K/mTOR signaling pathways, relevant downstream signaling network components, EGFR and VEGFR-related ligands, apoptosis (TUNEL), cell cycle control, and proliferation.
* To assess pre- and/or post-treatment tumor samples, when available, for DNA-based changes (e.g., EGFR [DNA] amplification, EGFR and EGFRvIII mutations, and mutations/deletions in the PTEN gene) relevant to the molecular biology in GBM.

OUTLINE: Patients receive oral erlotinib hydrochloride and sirolimus once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor tissue and blood sample collection periodically for pharmacological and biological studies. Samples are analyzed for concentrations of erlotinib hydrochloride and trough serum levels of sirolimus via HPLC, EGFR, EGFRvIII, PTEN and the phospho-specific antibodies associated with the MAPK and PI3K pathways via IHC, and EGFRvIII and sequencing of EGFR, PTEN and other critical genes via PCR, gene expression, and SNP analysis. Germline DNA will also be used to distinguish polymorphisms from somatic mutations in gene sequenced.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant glioma, including any of the following:
* Glioblastoma multiforme (GBM)
* Gliosarcoma (GS)
* Anaplastic astrocytoma (AA)
* Anaplastic oligodendroglioma (AO)
* Anaplastic mixed oligoastrocytomas (AMA)
* Malignant astrocytoma not otherwise specified (NOS)
* Prior low-grade glioma allowed provided there is histologic evidence of progression to a malignant glioma
* Must meet the following criteria for phase I:
* All types of malignant gliomas allowed
* No limitations on the number of relapses
* Must meet the following criteria for phase II:
* Only patients with GBM or GS are allowed
* Must be in first, second, or third relapse
* patients who had prior therapy (must include external beam radiotherapy) for a low-grade glioma that is considered standard, non-surgical treatment for a high-grade glioma, the surgical diagnosis of high-grade glioma will be considered the first relapse
* Must have shown unequivocal radiographic evidence for tumor progression by MRI or CT scan and have either measurable or evaluable disease
* Measurable disease is defined as bidimensionally measurable lesions with clearly defined margins by MRI scan
* Evaluable disease is defined as unidimensionally measurable lesions or masses with margins not clearly defined
* Karnofsky performance status ≥ 60%
* Life expectancy > 8 weeks
* Absolute neutrophil count ≥ 1,500/μL
* Platelets ≥ 100,000/μL
* Total bilirubin < 2.0 x upper limit of institutional normal (ULN)
* AST < 2.0 x ULN
* Creatinine < 1.5 x ULN
* Fasting serum triglycerides < 2.5 x ULN
* Fasting serum cholesterol < 350 mg/dL
* Women of child-bearing potential and men must agree to use adequate contraception (i.e., hormonal or barrier method of birth control) prior to study entry and for the duration of study participation
* Recovered from all toxicities associated with prior surgery, radiotherapy, or chemotherapy
* At least 1 week since prior surgery
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* At least 12 weeks since prior radiation therapy
* Must not receive any P450-enzyme-inducing anticonvulsants (EIAC) for at least 2 weeks prior to and during participation in this trial

Exclusion Criteria:

* Women who are pregnant or lactating
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib hydrochloride or sirolimus
* Uncontrolled intercurrent illness including, but not limited to, any of the following:
* Ongoing or active infection requiring IV antibiotics
* Symptomatic congestive heart failure
* Unstable angina pectoris
* Cardiac arrhythmia
* Hyperlipidemia (e.g., grade 3 or greater hypercholesterolemia or hypertriglyceridemia) not controlled with medication
* Psychiatric illness or social situations that would limit compliance with study requirements
* Disorders associated with significant immunocompromise (e.g., HIV or systemic lupus erythematosus [SLE])
* Patients with another primary malignancy that has required treatment other than surgery within the past year (except for nonmelanoma skin cancer or carcinoma in situ)
* Patients with the inability to comply with the protocol requirements in the opinion of the investigator including those who can not take oral medications
* Patients who are unable to undergo routine imaging evaluations with magnetic resonance imaging scans
* Prior EGFR-directed or mTOR-directed therapies including sirolimus or sirolimus analogs
* Patients taking concurrent immunosuppressive agents other than prescribed corticosteroids
* Concurrent antineoplastic or antitumor agents that are not part of the study therapy including chemotherapy, radiation therapy, immunotherapy, and hormonal anticancer therapy
* Blood products during cycle 1 unless a patient experiences hematologic DLT or if it is medically imperative to administer a transfusion
* Concurrent grapefruit or grapefruit juice
* Other concurrent investigational agents
* Receiving concurrent enzyme-inducing antiepileptic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-08; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To determine maximum tolerated dose and dose limiting toxicity of escalating doses of erlotinib in combination with sirolimus | day 28 of cycle 1

SECONDARY OUTCOMES:
To characterize the single-dose pharmacokinetic (PK) profile of erlotinib (in serum) and sirolimus (in whole blood) combination therapy in these patient populations | Day 1 of cycle 1
To characterize repeated-dose pharmacokinetic (PK) profile of erlotinib (in serum) and sirolimus (in whole blood) combination therapy in these patient populations | Day 28 of cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Timothy F. Cloughesy, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States